CLINICAL TRIAL: NCT03971500
Title: Comparison of 1-month Versus 12-month Dual Antiplatelet Therapy After Implantation of Drug-Eluting Stents Guided by Either Intravascular Ultrasound or Angiography in Patients With Acute Coronary Syndrome: The Prospective, Multicenter, Randomized, Placebo-controlled IVUS-ACS and ULTIMATE-DAPT Trials
Brief Title: 1-month vs 12-month DAPT for ACS Patients Who Underwent PCI Stratified by IVUS: IVUS-ACS and ULTIMATE-DAPT Trials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFH20190529
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Aspirin; Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1 randomization (first randomization) to either IVUS-guided DES implantation which will be the treatment group or Angio-guided DES implantation which will be the control group based on an online Clinical Research Data Management Platform. The initiation of the trial is defined as the time of randomization. After study subjects' enrollment and randomization, the study intervention will take place immediately. The follow-up visits for the primary TVF endpoint are scheduled at 1, 4, 6, and 12 months after the index procedure.
  Patients will undergo 1:1 randomization (second randomization) to either SAPT which will be the treatment group or DAPT which will be the control group based on an online Clinical Research Data Management Platform. The follow-up visits for the primary superiority bleeding endpoint and non-inferiority ischemic endpoint are scheduled at 3, 5, and 11 months after the second randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- IVUS-guidance (Experimental): In the IVUS-guided DES implantation group, optimal stent deployment criteria included: 1) the MLA in the stented segment is >5.0 mm^2, or 90% of the MLA at the distal reference segments; 2) plaque burden 5-mm proximal or distal to the stent edge is <55%; and 3) absence of >=Type B edge dissection. Further treatment will be required if any of those 3 criteria was not met.
  Interventions: Drug: AntiPlatelet therapy; Procedure: Percutaneous coronary intervention
- Angiography-guidance (Active Comparator): In the Angiography-guided DES implantation group, stent diameter and length will be selected by visual estimation with a stent/artery ratio of 1.1:1.0. Post-dilation with a noncompliant balloon (balloon/stent diameter=1.0:1.0) inflated at >18 atm will be performed for all lesions. Angiographic success is defined as Thrombolysis In Myocardial Infarction (TIMI) grade 3, residual stenosis <20%, and the absence of >Type B dissection.
  Interventions: Drug: AntiPlatelet therapy; Procedure: Percutaneous coronary intervention
- SAPT group (Experimental): Ticagrelor + aspirin for 1 month followed by ticagrelor plus matching placebo for an additional 11 months.
  Interventions: Drug: AntiPlatelet therapy; Procedure: Percutaneous coronary intervention
- DAPT group (Active Comparator): Ticagrelor + aspirin for 12 month.
  Interventions: Drug: AntiPlatelet therapy; Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Drug: AntiPlatelet therapy — AntiPlatelet therapy with ticagrelor + aspirin or ticagrelor alone.
  Other Names: ticagrelor, aspirin
Procedure: Percutaneous coronary intervention — PCI with DES implantation
  Other Names: PCI

SUMMARY:
Prospective, multicenter, randomized, double-blind, placebo-controlled trials.

DETAILED DESCRIPTION:
A total of 3486 subjects with ACS who met inclusion criteria and do not have any exclusion criterion will be randomized to IVUS- or Angiography-guidance group (first randomization). In the IVUS-guidance group, IVUS will be used to evaluate the lesion's specificity and to measure lesion length, landing zone, and reference vessel diameter prior-to stenting; and to assess stent expansion, extension, apposition, and possible complications after stent implantation. The IVUS- defined criteria for the optimal stent deployment included: 1) the minimal stent area (MSA) in the stented segment is >5.0 mm^2, or 90% of the MLA at the distal reference segments; 2) plaque burden 5-mm proximal or distal to the stent edge is <55%; and 3) absence of >Type B edge dissection. Further treatment will be required if stenting procedure is defined as suboptimal according to IVUS definition. IVUS will be not allowed to be used in the Angiography-guidance group.

Those patients who have had no death, STEMI, stroke, ST, TVR or major bleeding (BARC 3 or 5) within 30 days and have continued on aspirin and ticagrelor for 30 days without interruption for >48 hours will be randomized 1:1 to:

1. Ticagrelor plus+ matching placebo for an additional 11 months (SAPT group)
2. Ticagrelor plus aspirin (study drug) for an additional 11 months (DAPT group) Follow-up of all subjects will continue for 1 year with an option for additional follow-up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

Enrollment into the study will require meeting at least one of these clinical syndromes within 1 month.

* Unstable angina, defined as rest pain for 5-30 minutes or deteriorative exertional angina with either a) transient ST segment depression or elevation, or b) angiography showing a visually estimated diameter stenosis ≥90% or a ruptured plaque or thrombotic lesion
* Non-ST elevation myocardial infarction (NSTEMI), defined as positive troponin consistent with clinical syndrome.
* ST elevation MI (STEMI)

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Stroke within 3 months or any permanent neurologic deficit, and prior intracranial bleed, or any intracranial disease such as aneurysm or fistula
* Previous coronary artery bypass graft (CABG)
* Any planned surgery within 90 days
* Any reason why any antiplatelet therapy might need to be discontinued within 12 months
* Severe chronic kidney disease defined as an estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m^2
* Need for chronic oral anticoagulation (warfarin/coumadin or direct oral anticoagulants)
* Platelet count < 100,000 mm^3
* Contraindication to aspirin
* Contraindication to ticagrelor
* Liver cirrhosis
* Women of child-bearing potential
* Life expectancy < 1 year
* Any condition likely to interfere with study processes including medication compliance or follow-up visits (e.g. dementia, alcohol abuse, severe frailty, long distance to travel for follow-up visits, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3710 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 12 months
  The difference in TVF will be calculated from 0 month to 12 months between IVUS- and Angiography guidance groups.
Clinically-relevant bleeding | 11 months
  The difference in clinically-relevant bleeding (BARC ≥2) will be calculated from 1 month to 12 months between SAPT and DAPT groups.
Major adverse cardiovascular and cerebrovascular events (MACCE) | 11 months
  The difference in MACCE will be calculated from 1 month to 12 months between SAPT and DAPT groups.

SECONDARY OUTCOMES:
Net adverse clinical events (NACE) | 12 months
  The difference in NACE between IVUS- and Angiography guidance groups, or SAPT and DAPT groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Gao X, Kan J, Ge Z, Han L, Lu S, Tian N, Lin S, Lu Q, Wu X, Li Q, Liu Z, Chen Y, Qian X, Wang J, Chai D, Chen C, Li X, Gogas BD, Pan T, Shan S, Ye F, Chen SL. Intravascular Ultrasound Versus Angiography-Guided Drug-Eluting Stent Implantation: The ULTIMATE Trial. J Am Coll Cardiol. 2018 Dec 18;72(24):3126-3137. doi: 10.1016/j.jacc.2018.09.013. Epub 2018 Sep 24. PMID 30261237
- [Background] Ge Z, Gao XF, Kan J, Kong XQ, Zuo GF, Ye F, Tian NL, Lin S, Liu ZZ, Shao YB, He YQ, Wen SY, Yang Q, Xia Y, Wang ZZ, Xiao PX, Li F, Zeng HS, Yang S, Wang Y, Tao L, Gao DS, Qu H, Qian XS, Han YL, Chen F, Zhang JJ, Chen SL. Comparison of one-month versus twelve-month dual antiplatelet therapy after implantation of drug-eluting stents guided by either intravascular ultrasound or angiography in patients with acute coronary syndrome: rationale and design of prospective, multicenter, randomized, controlled IVUS-ACS and ULTIMATE-DAPT trial. Am Heart J. 2021 Jun;236:49-58. doi: 10.1016/j.ahj.2021.02.014. Epub 2021 Feb 20. PMID 33621541
- [Derived] Gao X, Kan J, Wu Z, Anjun M, Chen X, Chen J, Sheiban I, Mintz GS, Zhang JJ, Stone GW, Chen SL; IVUS-ACS Investigators. IVUS-Guided vs Angiography-Guided PCI in Patients With Diabetes With Acute Coronary Syndromes: The IVUS-ACS Trial. JACC Cardiovasc Interv. 2025 Feb 10;18(3):283-293. doi: 10.1016/j.jcin.2024.09.061. Epub 2024 Oct 28. PMID 39466211
- [Derived] Li X, Ge Z, Kan J, Anjum M, Xie P, Chen X, Khan HS, Guo X, Saghir T, Chen J, Gill BUA, Guo N, Sheiban I, Raza A, Wei Y, Chen F, Mintz GS, Zhang JJ, Stone GW, Chen SL; IVUS-ACS Investigators. Intravascular ultrasound-guided versus angiography-guided percutaneous coronary intervention in acute coronary syndromes (IVUS-ACS): a two-stage, multicentre, randomised trial. Lancet. 2024 May 11;403(10439):1855-1865. doi: 10.1016/S0140-6736(24)00282-4. Epub 2024 Apr 8. PMID 38604212
- [Derived] Ge Z, Kan J, Gao X, Raza A, Zhang JJ, Mohydin BS, Gao F, Shao Y, Wang Y, Zeng H, Li F, Khan HS, Mengal N, Cong H, Wang M, Chen L, Wei Y, Chen F, Stone GW, Chen SL; ULTIMATE-DAPT investigators. Ticagrelor alone versus ticagrelor plus aspirin from month 1 to month 12 after percutaneous coronary intervention in patients with acute coronary syndromes (ULTIMATE-DAPT): a randomised, placebo-controlled, double-blind clinical trial. Lancet. 2024 May 11;403(10439):1866-1878. doi: 10.1016/S0140-6736(24)00473-2. Epub 2024 Apr 7. PMID 38599220